CLINICAL TRIAL: NCT03791333
Title: A Multi-center Clinical Study on the Status of Trauma Evaluating Ability in Patients With Multiple Trauma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, wang tianbing, department of orthopaedic and trauma, Peking University People's Hospital
Other Study IDs: PUPH20181127
Record Dates: First submitted 2018-12-31; First posted 2019-01-02 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Multiple Trauma/Injuries
MeSH Terms: conditions — Multiple Trauma; Wounds and Injuries | interventions — Injury Severity Score

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- multi trauma patients group
  Interventions: Other: injury severity score

INTERVENTIONS:
Other: injury severity score — injury severity score of multi trauma patients

SUMMARY:
Trauma is a major medical and public health problem facing all countries in the world today. Trauma is the leading cause of death worldwide for people under 45 years of age, and more than 5 million people die each year from severe trauma. According to the "China Injury Prevention Report" issued by the Ministry of Health in August 2007, about 200 million injuries occur annually in China, with 700,000 to 750,000 deaths, accounting for about 9% of the total number of deaths. Serious trauma has the characteristics of high mortality and disability rate, and often affects the main groups of young and middle-aged people of social labor force. It has a tremendous impact on social and economic development, and has brought a heavy burden to society and families. The treatment of severe trauma is extremely important, and its treatment process needs a standardized model. In many links of trauma treatment, accurate assessment of injury is the precondition of classification and grading of diagnosis and treatment, and also provides a good basis for the follow-up standardized treatment of patients. The accuracy and consistency of injury assessment are also the reflection of diagnosis and treatment ability. ISS score is an evaluation method for severe trauma and multiple trauma patients. It has been used by emergency personnel for a long time. It also plays a very good auxiliary role in the evaluation and treatment of patients'injuries. However, there are still many problems in the clinical use of ISS scores: 1. Some hospitals do not attach importance to the application of ISS scores, and do not fully understand the scoring method; 2. Low frequency of use, inaccurate grasp of the method; 3. Three-level physicians have different valuations of ISS scores for the same kind of trauma; 4. Use AIS scoring table to calculate. It takes a long time to calculate the ISS score, which affects the normal first aid efficiency. To this end, our research team designed a questionnaire on the use of ISS score. The main purpose of the questionnaire is to assess and register the severity of injury in multiple trauma patients to understand the current use and proficiency of ISS score system by Chinese trauma surgeons, the difference of ISS score between three-level doctors and the same patient, and ISS score. The consistency between the software and AIS scoring table and the scoring time of the two methods are also discussed. This study hopes that through this survey, we can understand the current situation of the application of the scoring system in Chinese hospitals, in order to promote the standardization of severe trauma assessment and promote the use of the evaluation system in hospitals throughout the country, so as to provide optimized trauma treatment process for trauma patients.

DETAILED DESCRIPTION:
1. Research Background and Basis for Project Establishment* Trauma is a major medical and public health problem facing all countries in the world today. Trauma is the leading cause of death worldwide for people under 45 years of age, and more than 5 million people die each year from severe trauma. According to the "China Injury Prevention Report" issued by the Ministry of Health in August 2007, about 200 million injuries occur annually in China, with 700,000 to 750,000 deaths, accounting for about 9% of the total number of deaths. Serious trauma has the characteristics of high mortality and disability rate, and often affects the main groups of young and middle-aged people of social labor force. It has a tremendous impact on social and economic development, and has brought a heavy burden to society and families. The treatment of severe trauma is extremely important, and its treatment process needs a standardized model. In many links of trauma treatment, accurate assessment of injury is the precondition of classification and grading of diagnosis and treatment, and also provides a good basis for the follow-up standardized treatment of patients. The accuracy and consistency of injury assessment are also the reflection of diagnosis and treatment ability. ISS score is an evaluation method for severe trauma and multiple trauma patients. It has been used by emergency personnel for a long time. It also plays a very good auxiliary role in the evaluation and treatment of patients'injuries. However, there are still many problems in the assessment of severe trauma in various parts of China. It is difficult to adapt to the needs of the current medical and health system reform and to meet the needs of the society for the assessment of severe trauma. In the clinical use of ISS scoring, the main problems are as follows: 1. Some hospitals do not attach importance to the application of ISS scoring, and do not fully understand the scoring method; 2. The use of low frequency, inaccurate grasp of the method; 3. Three-level physicians have different evaluation of ISS scoring for the same kind of trauma; 4. Applying AIS scoring table to calculate ISS scoring. It takes a long time to share the time, which affects the normal first aid efficiency.
2. Research purposes * By assessing and registering the severity of multiple trauma patients, we can understand and improve the ability of different hospitals and doctors at different levels in different regions to assess the severity of multiple trauma patients, and promote the use of ISS scoring system in national trauma centers. In order to improve the level of understanding of multiple trauma patients and lay a foundation for the establishment of scientific classification and sorting and treatment system.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age not less than 18 years old; 2. Multiple trauma patients; 3. Complete auxiliary examination data of various trauma sites.

Exclusion Criteria:

* Patients who died on the spot or came to hospital; pregnant and lying-in women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple injuries who visited our research centers
Sampling Method: Non-Probability Sample
Enrollment: 3600 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
ISS score of third-level surgeons for the same patient | 3 years
  ISS score of third-level surgeons for the same patient
Scoring time | 3 years
  Scoring spending time

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kirkpatrick JR, Youmans RL. Trauma index. An aide in the evaluation of injury victims. J Trauma. 1971 Aug;11(8):711-4. No abstract available. PMID 5565650
- [Background] Koehler JJ, Baer LJ, Malafa SA, Meindertsma MS, Navitskas NR, Huizenga JE. Prehospital Index: a scoring system for field triage of trauma victims. Ann Emerg Med. 1986 Feb;15(2):178-82. doi: 10.1016/s0196-0644(86)80016-6. PMID 3946860
- [Background] Jennett B. The Glasgow Coma Scale: History and current practice. Trauma, 2002, 4(2):91-103.
- [Background] Baker SP, O'Neill B, Haddon W Jr, Long WB. The injury severity score: a method for describing patients with multiple injuries and evaluating emergency care. J Trauma. 1974 Mar;14(3):187-96. No abstract available. PMID 4814394